CLINICAL TRIAL: NCT05146024
Title: WayToServe Plus: In-service Professional Development Component to Improve Responsible Alcohol Service Ph I
Brief Title: WayToServePlus: Improving Responsible Alcohol Service Ph I
Status: Completed | Type: Observational
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: Pacific Institute for Research and Evaluation (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0332; 1R44AA029364-01 (NIH)
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Driving While Intoxicated
Keywords: Alcohol Use; Prevention
MeSH Terms: conditions — Driving Under the Influence; Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Formative Research: Alcohol-serving establishment owners, managers, and servers in New Mexico and Washington State.
  Interventions: Behavioral: Way To Serve Plus: Improving Responsible Alcohol Service

INTERVENTIONS:
Behavioral: Way To Serve Plus: Improving Responsible Alcohol Service — Improving responsible alcohol service of owners, managers, and employees of alcohol-serving establishments by developing professional development components to enhance their responsible beverage service skills.

SUMMARY:
Responsible beverage service (RBS) training for alcohol servers is a promising intervention for reducing driving while intoxicated (DWI) by alcohol. Training, certification, and in-service contact improves professionalism and effectiveness of prevention interventions delivered by community members such as alcohol servers. This SBIR Fast-track project will develop and test an in-service professional development component to the WayToServe® online RBS training to improve the effectiveness of RBS training in order to make further gains in reducing problem alcohol behavior in communities.

DETAILED DESCRIPTION:
Among the interventions targeting driving while intoxicated (DWI) by alcohol, Responsible Beverage Service (RBS) training of alcohol servers has shown promise. RBS training is currently required or incentivized by 36 U.S. states and California will require it starting in 2022. Our team has shown that an online RBS training, named WayToServe®, was effective in two randomized trials. These results filled a gap in the literature on RBS training that is limited by the lack of randomized trials, poor measurement of training implementation, and almost exclusive focus on live training when online training predominates. The goal of this SBIR Fast-track research is to develop and test an in-service professional development component for alcohol servers trained by WayToServe to improve its effectiveness. It is intended to motivate servers to implement the RBS skills in the face of common barriers, provide support for RBS actions from a "community" of alcohol servers, and prevent natural degradation of skills over time. Rationale for this product is provided by past research showing that training, certification, and in-service contact improves professionalism and efficacy of community prevention interventions. Scientific premise is provided by the positive results of our trials on the WayToServe® training. The in-service component will be delivered through the WayToServe Facebook page that currently is "followed" by over 20,000 alcohol servers trained by WayToServe. The specific aims of Phase I are to: 1) develop content of in-service professional development on RBS skills with a) premises owners/ managers interviews and b) alcohol servers in New Mexico and Washington State trained by the WayToServe online RBS training through focus group discussions; 2) produce a prototype WayToServe Plus in-service professional development component in flowcharts and an initial library of Facebook posts, including text, graphics, and interactive elements and evaluate it for acceptability, usability, and engagement in focus groups and field pilot trial with alcohol servers in New Mexico and Washington State trained by the WayToServe online RBS training, and 3) determine feasibility of WayToServe Plus in-service professional development component and develop evaluation plans for Phase II research. Milestones will be an EAB-approved Phase I research plans and development of the content outline and WayToServe Plus prototype, evaluation of WayToServe Plus prototype, and feasibility assessment of the WayToServe Plus in-service professional development component. Phase II specific aims will achieve the milestones of full production of WayToServe Plus and a randomized trial testing its effectiveness by: 4) producing the full WayToServe Plus in-service professional development component and 5) conducting a randomized trial with 160 alcohol premises in New Mexico and Washington State evaluating effectiveness of WayToServe Plus on refusal of sales to PiP (primary outcome). The SBIR research is innovative as WayToServe Plus will be the first continuous in-service professional development for RBS and will increase the WayToServe training's effectiveness and commercial advantage with alcohol servers and corporate clients.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* Own/manage a licensed premises or be an alcohol server (waitress, waiter or bartender)
* Have completed the WayToServe responsible beverage service training (Phase I only)
* Be proficient in English
* Consent to participate

Exclusion Criteria:

* Have a family/household member already participating in project
* Younger than 19 years old (18 and younger cannot legally serve alcohol in either state)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Owners, managers, and employees of alcohol-serving establishments in New Mexico and Washington State.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Formative Research | Baseline Only
  Focus Groups, Semi-structured Interviews, Field Pilot Test

CONTACTS AND LOCATIONS:
Overall Officials: David Buller, PHD, Principal Investigator — Klein Buendel, Inc.; Gill Woodall, PhD, Principal Investigator — Klein Buendel, Inc.
Locations (2):
- United States (2):
  - Pacific Institute for Research and Evaluation, Berkeley, California
  - Klein Buendel, Inc., Golden, Colorado